CLINICAL TRIAL: NCT02718430
Title: VXM01 Phase I Study in Patients With Metastatic Colorectal Cancer With Liver Metastasis Under Second or Third Line Therapy to Examine Safety, Efficacy, and Immune Biomarkers After Treatment With VXM01
Brief Title: VXM01 Phase I Study in Patients With Metastatic Colorectal Cancer With Liver Metastasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaximm GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VXM01-03-DE
Record Dates: First submitted 2016-03-16; First posted 2016-03-24 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VXM01 (Experimental): VXM01 10E6 or 10E7 CFU
  Interventions: Drug: VXM01

INTERVENTIONS:
Drug: VXM01 — Oral immunotherapy targeting VEGFR2

SUMMARY:
Phase I study in patients with metastatic colorectal cancer with liver metastasis under second or third line therapy to examine safety, efficacy, and immune biomarkers after treatment with VXM01

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent, including liver metastasis biopsy, signed and dated
2. Histologically or cytologically confirmed colorectal cancer, excluding primary tumors of appendiceal origin (participants are eligible to enroll irrespective of Kirsten rat sarcoma viral oncogene homolog (KRAS) mutation status)
3. Male or female patients who must be post-menopausal for at least 2 years or surgically sterile.
4. Confirmed metastatic colorectal cancer (Stage IV)
5. Presence of non-resectable liver metastasis

   * Accessibility of liver metastasis appropriate for biopsy sampling
   * Adequate coagulation parameters including platelet count ≥100,000/mm3
   * Absence of concomitant medication which could represent a contraindication for biopsy (e.g., anti-platelet drugs including aspirin, ticlopidine, clopidogrel, IIb/IIIa receptor antagonists, non-steroidal anti-inflammatory drugs [NSAIDs], and vitamin K antagonist anticoagulants)
6. The participant has received first-line irinotecan- or oxaliplatin-based therapy without or in combination with a targeted antibody for metastatic disease and a) Experienced radiographic disease progression during first-line therapy, or b) Experienced radiographic disease progression ≤ 6 months after the last dose of first-line therapy, or c) Discontinued part or all of first-line therapy due to toxicity and experienced radiographic disease progression ≤ 6 months after the last dose of first-line therapy
7. Receipt of no more than 3 prior systemic therapy regimen for metastatic disease
8. Measurable or non-measurable disease based on the Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v. 1.1)
9. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
10. Life expectancy > 3 months
11. Adequate renal, hepatic, and bone marrow function
12. Leukocytes ≥4.0 x 109 / L
13. Absolute neutrophil count (ANC) > 1,500/mm3
14. Platelet count ≥ 100,000/mm3
15. Hemoglobin ≥ 9 g/dL (can be post-transfusion)
16. International normalized ratio (INR) ≤ 1.5
17. Activated partial thromboplastin time (aPTT) ≤ 1.5 times upper limit of normal (ULN)
18. Bilirubin ≤ 1.5 times ULN
19. ALT and AST ≤ 2.5 times ULN
20. Creatinine ≤ 2.0 mg/dL
21. Proteinuria ≤ 1+ by urine dipstick OR ≤ 1 g by 24-hour urine collection
22. Patients who are able to understand the nature and purpose of the study including possible risks, willing to comply with the requirements, and to provide their written informed consent to participate in the study

Exclusion Criteria:

1. Concomitant treatment with anti-angiogenic therapy before progression of disease
2. Treatment in any other clinical trial within 30 days before screening.
3. Gastric bypass
4. Ileostoma
5. Other anatomical change of the gastrointestinal tract, interfering with gastrointestinal passage, except colostoma or colon bypass
6. Untreated CNS metastases. Participants with treated brain metastases are eligible if they are clinically stable with regard to neurologic function, off steroids after cranial irradiation ending at least 2 weeks prior to randomization, or after surgical resection performed at least 28 days prior to randomization. No evidence of Grade greater than or equal to 1 CNS hemorrhage based on pretreatment Magnetic Resonance Imaging (MRI) or intravenous (IV) contrast CT scan
7. Significant traumatic injury or surgery within the past 4 weeks
8. Cerebrovascular accident, transient ischemic attack, or subarachnoid hemorrhage within the past 6 months
9. Other malignancies within the past 5 years except for adequately treated carcinoma in situ of the cervix, and/or basal cell skin cancer, and/or early endometrial carcinoma
10. Pre-existing sensory or motor neuropathy ≥ grade 2
11. History or evidence of CNS disease (e.g., uncontrolled seizures) by neurological examination unless adequately treated with standard medical therapy
12. History or evidence of thrombotic or hemorrhagic disorders, including intracranial hemorrhage
13. Uncontrolled hypertension (i.e., blood pressure > 160/100 mm Hg)
14. Clinically significant cardiovascular disease, including any of the following:

    * Myocardial infarction or unstable angina within the past 6 months
    * New York Heart Association class III-IV congestive heart failure
    * Poorly controlled cardiac arrhythmia despite medication, except rate controlled atrial fibrillation
15. Peripheral vascular disease ≥ grade 3 (i.e., symptomatic and interfering with activities of daily living requiring repair or revision)
16. Positive for anti-typhoid IgG/IgM antibodies according to the onsite test on Day 0
17. Hemoptysis within 6 months before randomization
18. Esophageal varices
19. Upper or lower gastrointestinal bleeding within 6 months before randomization
20. Non-healing wound, incomplete wound healing, bone fracture or any history of gastrointestinal ulcers within three years before inclusion, or positive gastroscopy within 3 months before inclusion
21. Gastrointestinal fistula
22. Thrombolysis therapy within 4 weeks before randomization
23. Presence of any acute or chronic systemic infection
24. Major surgical procedures, or open biopsy within 4 weeks before randomization
25. Chronic concurrent therapy within 2 weeks before and during the initial treatment period (Day 1 to Day 7):

    * Corticosteroids (except steroids for adrenal failure or emesis prophylaxis up to 4 mg daily dose) or immunosuppressive agents
    * Antibiotics
    * Bevacizumab or any other anti-angiogenic treatment
26. Known multi-drug resistant gram-negative bacteria
27. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the study results or render the patient at high risk for treatment complications
28. Women of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-02; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability taking into account treatment-limiting toxicities (TLTs) | 18 months
  AEs listed together with information on onset, duration, severity, seriousness, relationship to the study drug, relationship to chemotherapy and to the underlying disease, outcome, and action taken. Frequency tables by System Organ Class and preferred term.

SECONDARY OUTCOMES:
Immune Response by Enzme Linked Immuno Spot (ELISpot) | 18 months
  Patient-individual VEGFR-2 specific T-cell responses determined by ELISpot using cryopreserved peripheral blood mononuclear cells (PBMC)
Immune biomarker by tumor tissue immunohistochemistry staining | 66 days
  Immune biomarker including T-cell infiltration, Treg, myeloid derived suppressor cells (MDSC) by tumor tissue immunohistochemistry staining
Tumor vasculature by tumor tissue immunohistochemistry staining | 66 days
Serum biomarker Response by Enzyme Linked Immuno Sorbent Assay (ELISA) | 18 months
  Serum VEGF A and collagen IV measured by ELISA
Clinical Response including tumor staging according to the response criteria in solid tumors (RECIST) | 18 months
  Tumor staging according to the response criteria in solid tumors (RECIST) and investigation of the primary tumor and metastasis, e.g., determination of primary tumor size, number and size of metastasis.
Biodistribution and shedding of VXM01 | 10 days
  Bacterial vector tissue biodistribution, persistence, and shedding of viable Ty21a bacteria (VXM01) determined by cultivation of stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Gruellich, MD, Principal Investigator — National Center of Tumor Diseases Heidelberg
Locations (1):
- National Center of Tumor Diseases, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Yes